CLINICAL TRIAL: NCT00581139
Title: Psychological Influences on Postoperative Recovery
Acronym: NIH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Zeev Kain, Professor, University of California, Irvine
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 9801009972 [2008-6723]; R01HD037007-01 (NIH)
Record Dates: First submitted 2007-12-18; First posted 2007-12-27 (Estimated); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Care, Postoperative; Pain, Postoperative; Surgical Procedures, Operative; Otorhinolaryngologic Surgical Procedures; Tonsillectomy; Adenoidectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Allied Health Personnel; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator)
  Interventions: Behavioral: Preoperative Preparation Program (Child Life Specialist)
- 2 (Active Comparator)
  Interventions: Drug: Midazolam
- 3 (Active Comparator)
  Interventions: Behavioral: Parental Presence during Induction of Anesthesia
- 4 (Active Comparator)
  Interventions: Other: PPIA preparation program PLUS Midazolam premedication

INTERVENTIONS:
Behavioral: Preoperative Preparation Program (Child Life Specialist) — This group will receive the standard preoperative visit to the hospital with Child Life intervention
  Arms: 1
Drug: Midazolam — 0.5 mg/kg oral midazolam
  Other Names: Versed
  Arms: 2
Behavioral: Parental Presence during Induction of Anesthesia — One parent will be present during induction of anesthesia of the child. The parent will be accompanied out of the OR by a nurse once the induction is completed. These parents will have completed a parent preparation program.
  Other Names: PPIA Preparation Program
  Arms: 3
Other: PPIA preparation program PLUS Midazolam premedication — Subjects in this group will receive both interventions 2 and 3.
  Arms: 4

SUMMARY:
The primary hypothesis tested in this project is that the preoperative behavioral stress response predicts postoperative behavioral and clinical recovery of children undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient tonsillectomy or tonsils/adenoids
* ASA I, II

Exclusion Criteria:

* Developmental delay
* ASA III-IV
* Psychotropic medication
* Meds which interfere with metabolism of midazolam
* 36 weeks gestation

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 241 (Actual)
Dates: Start 2003-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeev N Kain, MD, MBA, Principal Investigator — Yale University Department of Anesthesiology
Locations (1):
- Yale University Department of Anesthesiology, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between 2003 and 2009 at the Yale Children's Hospital.
Pre-assignment Details: All enrolled participants were assigned to one of the four groups.
Groups:
- Standard of Care: Preoperative Preparation Program (Child Life Specialist) : This group will receive the standard preoperative visit to the hospital with Child Life intervention
- Pre-medication: Midazolam : 0.5 mg/kg oral midazolam
- Parental Presence During Induction of Anesthesia: Parental Presence during Induction of Anesthesia : One parent will be present during induction of anesthesia of the child. The parent will be accompanied out of the OR by a nurse once the induction is completed. These parents will have completed a parent preparation program.
- Parental Presence During Induction of Anesthesia PLUS Premedic: PPIA preparation program PLUS Midazolam premedication : Subjects in this group will receive both interventions 2 and 3.
Period: Overall Study
Arm/Group | Standard of Care | Pre-medication | Parental Presence During Induction of Anesthesia | Parental Presence During Induction of Anesthesia PLUS Premedic
Started | 61 | 68 | 54 | 58
Completed | 61 | 68 | 54 | 58
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Pre-medication | Parental Presence During Induction of Anesthesia | Parental Presence During Induction of Anesthesia PLUS Premedic | Total
Number analyzed (Participants) | 57 | 66 | 54 | 56 | 233
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.59 (2.578) | 7.56 (6.48) | 6.57 (2.57) | 6.74 (2.50) | 6.96 (4.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 38 | 31 | 33 | 127
  Male | 32 | 28 | 23 | 23 | 106

OUTCOME MEASURES:

1. Primary Outcome: Modified Yale Preoperative Anxiety Scale
Description: The Modified Yale Preoperative Anxiety Scale (mYPAS) is the current "criterion standard" for assessing child anxiety during induction of anesthesia and has been used in >100 studies. This observational instrument covers 5 items and is typically administered at 4 perioperative time points. Minimum value is 23.33 and maximum value is 100. Scores below 30 are considered low anxiety. Score of 30 or more is considered high anxiety.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: Score on mYPAS scale
Arm/Group | Standard of Care | Pre-medication | Parental Presence During Induction of Anesthesia | Parental Presence During Induction of Anesthesia PLUS Premedic
Number analyzed (Participants) | 56 | 60 | 54 | 55
Score on mYPAS scale | 41.59 (22.18) | 37.44 (21.80) | 46.17 (24.10) | 33.65 (15.23)
Statistical Analysis 1: Comparison: Standard of Care vs Pre-medication vs Parental Presence During Induction of Anesthesia vs Parental Presence During Induction of Anesthesia PLUS Premedic; Test type: Superiority; p = .02, ANOVA

2. Primary Outcome: Percentage of Children Not Exhibiting Negative Behaviors, Fear, or Anxiety (Perfect Induction, 0)
Description: A total score is the number of categories checked (1-10). A perfect induction is when a patient does not exhibit negative behaviors, fear, or anxiety. A perfect score would be 0.
  icc 1 = Crying, tears in eyes
  icc 2 = Turns head away from mask
  icc 3 = Verbal refusal, says "no"
  icc 4 = Verbalization indicating fear or worry, "Where's mommy?" or "Will it hurt?"
  icc 5 = Pushes mask away with hands, pushes nurse/anesthesiologist with hands/feet
  icc 6 = Covers mouth/nose with hands/arms or buries face
  icc 7 = Hysterical crying, may scream
  icc8 = Kicks/flails legs/arms, arches back, and/or general struggling
  icc9 = Requires physical restraint
  icc10 = Complete passivity either rigid or limp
  icc 0 = Perfect induction
Time Frame: Induction, up to 10 minutes
Population: The discrepancy noted in the analysis population is due to missing data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Standard of Care | Pre-medication | Parental Presence During Induction of Anesthesia | Parental Presence During Induction of Anesthesia PLUS Premedic
Number analyzed (Participants) | 56 | 60 | 54 | 55
Percentage of Participants | 68 | 83 | 62 | 86

3. Primary Outcome: Percent of Children Crying During Induction
Description: Children who were crying/ had tears in their eyes during induction.
Time Frame: Induction, up to 10 minutes
Population: The discrepancy noted in the analysis population is due to missing data
Measure: Number; unit: Percentage of Participants
Arm/Group | Standard of Care | Pre-medication | Parental Presence During Induction of Anesthesia | Parental Presence During Induction of Anesthesia PLUS Premedic
Number analyzed (Participants) | 56 | 60 | 54 | 55
Percentage of Participants | 32 | 17 | 38 | 14
Statistical Analysis 1: Comparison: Standard of Care vs Pre-medication vs Parental Presence During Induction of Anesthesia vs Parental Presence During Induction of Anesthesia PLUS Premedic; Test type: Superiority; p = .01, Chi-squared

4. Primary Outcome: Percentage of Children Arriving to PACU Awake
Description: Whether child arrived to PACU awake Emergence of 1 // whether child arrived to PACU awake
Time Frame: Arrival at PACU, after surgery up to 20 minutes
Population: The discrepancy noted in the analysis population is due to missing data
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care | Pre-medication | Parental Presence During Induction of Anesthesia | Parental Presence During Induction of Anesthesia PLUS Premedic
Number analyzed (Participants) | 56 | 60 | 54 | 55
Percentage of participants | 55 | 32 | 32 | 33
Statistical Analysis 1: Comparison: Standard of Care vs Pre-medication vs Parental Presence During Induction of Anesthesia vs Parental Presence During Induction of Anesthesia PLUS Premedic; Test type: Superiority; p = .01, Chi-squared

5. Primary Outcome: Percentage of Children Arriving to PACU in Deep Sleep
Description: Whether child arrived to PACU awake Emergence of 2 // whether child arrived to PACU in deep sleep
Time Frame: Arrival at PACU, after surgery up to 20 minutes
Population: The discrepancy noted in the analysis population is due to missing data
Measure: Number; unit: Percentage of Participants
Arm/Group | Standard of Care | Pre-medication | Parental Presence During Induction of Anesthesia | Parental Presence During Induction of Anesthesia PLUS Premedic
Number analyzed (Participants) | 56 | 60 | 54 | 55
Percentage of Participants | 45 | 68 | 46 | 67
Statistical Analysis 1: Comparison: Standard of Care vs Pre-medication vs Parental Presence During Induction of Anesthesia vs Parental Presence During Induction of Anesthesia PLUS Premedic; Test type: Superiority; p = .01, Chi-squared

6. Primary Outcome: Post Anesthesia Care Unit (PACU) IV Fluid
Description: Total IV fluid per kg in PACU
Time Frame: Post Anesthesia Care Unit up to 2 hours
Population: The discrepancy noted in the analysis population is due to missing data
Measure: Mean (Standard Deviation); unit: mL/Kg
Arm/Group | Standard of Care | Pre-medication | Parental Presence During Induction of Anesthesia | Parental Presence During Induction of Anesthesia PLUS Premedic
Number analyzed (Participants) | 32 | 38 | 54 | 55
mL/Kg | 13.18 (8.39) | 16.85 (9.76) | 18.78 (11.44) | 22.21 (14.80)
Statistical Analysis 1: Comparison: Standard of Care vs Pre-medication vs Parental Presence During Induction of Anesthesia vs Parental Presence During Induction of Anesthesia PLUS Premedic; Test type: Superiority; p = .02, ANOVA

7. Primary Outcome: Visual Analogue Pain Scale (VAS) 24 Hour After Surgery
Description: Parent-ranted child pain on the Visual Analogue Scale. The VAS for pain is a unidimensional measure of pain presented in a horizontal line from 0-100. A higher score indicates greater pain intensity.
  0-4= no pain/anxiety, 5-44= mild pain/anxiety, 45-74 = moderate pain/anxiety, 75-100 = severe pain/anxiety.
Time Frame: 24 Hours after surgery
Population: The discrepancy noted in the analysis population is due to missing data
Measure: Mean (Standard Deviation); unit: Score on Visual Analogue Scale
Arm/Group | Standard of Care | Pre-medication | Parental Presence During Induction of Anesthesia | Parental Presence During Induction of Anesthesia PLUS Premedic
Number analyzed (Participants) | 32 | 36 | 54 | 55
Score on Visual Analogue Scale | 34.13 (21.98) | 35.93 (23.35) | 38.30 (24.30) | 47.02 (24.53)
Statistical Analysis 1: Comparison: Standard of Care vs Pre-medication vs Parental Presence During Induction of Anesthesia vs Parental Presence During Induction of Anesthesia PLUS Premedic; Test type: Superiority; p = .04, ANOVA

8. Primary Outcome: Heart Rate in the General Clinical Research Unit (GCRC)
Description: Heart rate was measured in the GCRC by the nurse hours 0 through 6 after Surgery
Time Frame: Hour 0-6 after surgery
Population: The discrepancy noted in the analysis population is due to missing data
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Standard of Care | Pre-medication | Parental Presence During Induction of Anesthesia | Parental Presence During Induction of Anesthesia PLUS Premedic
Number analyzed (Participants) | 32 | 38 | 54 | 55
beats per minute | 96.75 (17.99) | 95.13 (18.96) | 97.39 (18.32) | 104.55 (18.45)
Statistical Analysis 1: Comparison: Standard of Care vs Pre-medication vs Parental Presence During Induction of Anesthesia vs Parental Presence During Induction of Anesthesia PLUS Premedic; Test type: Superiority; p = .04, ANOVA

ADVERSE EVENTS:
Time Frame: 2-Weeks
Description: Use of standard questionnaires
Arm/Group | Standard of Care | Pre-medication | Parental Presence During Induction of Anesthesia | Parental Presence During Induction of Anesthesia PLUS Premedic
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/68 | 0/54 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/68 | 0/54 | 0/58
Other Adverse Events (participants affected / at risk) | 0/61 | 0/68 | 0/54 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No